CLINICAL TRIAL: NCT06693596
Title: Masses in Young Patients - International Ovarian Tumour Analysis: Prospective Validation and Comparison of Simple Rules, Benign Descriptors and ADNEX Models for Discrimination Between Benign and Malignant Adnexal Masses in Young Girls and Adolescents MY-IOTA
Brief Title: Masses in Young Patients - International Ovarian Tumour Analysis (MY-IOTA)
Acronym: MY-IOTA
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S68104
Record Dates: First submitted 2024-02-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-02

CONDITIONS: Adnexal Mass; Adnexal Tumor; Adnexal Cyst; Adnexal Masses in Young Girls and Adolescents
Keywords: IOTA; ovarian mass; benign; malignant; Young patients
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Surgical management: Patients aged ≤ 20 years of age recommended for surgery at that visit due to a suspicion of malignancy or pain.
  Interventions: Procedure: Group 1: Surgical management
- Group 2: Conservative management (follow-up): Patients aged ≤ 20 not recommended for surgery due to suspicion of malignancy/complications, for which subjective impression was benign for all visits, and for which the tumour was still present at the next visit.
  Interventions: Diagnostic Test: Group 2: Conservative management (follow-up)

INTERVENTIONS:
Diagnostic Test: Group 2: Conservative management (follow-up) — A standardised transabdominal examination is performed, including color or power Doppler examination. Transvaginal ultrasonography can be performed in sexually active adolescents with consent. Transrectal examination is also acceptable for younger patients who are not sexually active. All the variables required for the Simple Rules, simple descriptors and ADNEX model are assessed.
  Before entering ultrasound information about the tumour and getting model results, the ultrasound examiner' s diagnosis (benign, borderline, malignant; specific diagnosis) based on subjective assessment is recorded. Results based on Simple Rules, simple descriptors and ADNEX model are documented as well.
  If the adnexal mass is seen and if the decision is to manage the adnexal mass conservatively, the patient will be re-scanned at 6 weeks (maximal range 6-8 weeks), 3 months (+/- 2 weeks) and 12 months (maximal range 10-14 months)
  Other Names: Ultrasound Assessment
  Groups: Group 2: Conservative management (follow-up)
Procedure: Group 1: Surgical management — A standardised transabdominal examination is performed, including color or power Doppler examination. Transvaginal ultrasonography can be performed in sexually active adolescents with consent. Transrectal examination is also acceptable for younger patients who are not sexually active. All the variables required for the Simple Rules, simple descriptors and ADNEX model are assessed.
  Before entering ultrasound information about the tumour and getting model results, the ultrasound examiner' s diagnosis (benign, borderline, malignant; specific diagnosis) based on subjective assessment is recorded. Results based on Simple Rules, simple descriptors and ADNEX model are documented as well.
  If the patient requires surgery, no further ultrasound scans will be required.
  Other Names: Surgery
  Groups: Group 1: Surgical management

SUMMARY:
This multicenter observational study aims to validate the IOTA Simple Rules, Benign Descriptors, and ADNEX model in a cohort of patients equal or under the age of 20. Moreover, the study aims to evaluate the diagnostic accuracy of subjective assessment by ultrasound and to analyze the rate of complications in patients treated conservatively.

DETAILED DESCRIPTION:
Ovarian masses are uncommon in children, with an estimated annual incidence of 2.6/100,000. They are most identified in the neonatal period or around the time of menarche. Most ovarian cysts are benign and 55-70% of which are mature cystic teratomas. In most cases, patients are asymptomatic and the ovarian lesions are incidentally detected through ultrasound examinations. However, up to 15% of cases may involve abdominal pain and torsion. Furthermore, despite the low incidence of ovarian cancer (less than 1% of all pediatric cancers), the possibility of malignant tumor must be addressed.

In 2018, a national survey of pediatric surgeons in the UK revealed significant variability in the strategies employed for investigating and surgically managing adnexal lesions in children and adolescents. Although there is a spread consensus that ultrasound indices are useful for distinguishing between benign and malignant lesions in pediatric patient, the evidence available for this specific population is limited and it lacks comprehensive data from large cohorts. Moreover, existing models developed by the International Ovarian Tumor Analysis (IOTA) group, such as the Simple Rules, Benign Descriptors, and ADNEX model, have not been validated in this younger population. Additionally, it is still unclear if these tools remain validated with a transabdominal approach, primarily used for children and non-sexually active adolescents.

The primary objective of this prospective study is therefore to assess the performance of these existing ultrasonography-based risk tools in discriminating between benign and malignant adnexal masses in neonates, young girls and adolescents using transabdominal and/or transvaginal ultrasound.

Secondary aims are the diagnostic accuracy of subjective assessment by ultrasound, the understanding of the natural history of adnexal masses at 6-8 weeks, 3 months, and 12 months and the assessment of the complications rate (such as rupture, torsion, or malignancy) in patients treated conservatively.

Final outcome will be based on pathology in patients who undergo surgery and on pattern recognition, i.e. subjective assessment of ultrasound examiner, in patients managed conservatively for masses where morphology remains unchanged during follow-up.

The study will be conducted over a minimum of two years. We anticipate recruiting 1000 surgically managed masses over a 24-month period.

ELIGIBILITY:
• Inclusion Criteria:

All newly diagnosed adnexal masses identified in a girl or adolescent aged 20 or under.

• Exclusion Criteria:

Participants eligible for this study must not meet any of the following criteria:

* Non-adnexal masses e.g. peritoneal inclusion cysts (where diagnosis is certain) and peritoneal carcinomatosis with no adnexal mass;
* The denial or withdrawal of written informed consent.
* Pregnancy at any timepoint during the study period
* In premenarchal participants: follicle measuring <10mm

Ages: 0 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients under 18 years of age newly diagnosed with adnexal masses in the study centre (UZ Leuven) or in one of the other affiliated hospitals and who underwent both conservative and surgical management.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2026-07-21 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Estimation of the ability of the ADNEX model without CA125 to discriminate between benign and malignant adnexal masses when detected in patients aged 20 or under (AUC) | Outcome based on histology for group 1 assessed at 12 months after recruitment or no sign of malignancy during the ultrasound follow-up for group 2 assessed up to 12 months after recruitment.
  Area under the receiver operating characteristic curve (AUC). This will be done using the estimated probability of malignancy, which equals 1 minus the estimated probability of a benign tumor. 95% confidence intervals provided. Analysis will be done twice: for subgroup 1 and for subgroups 1 and 2 combined.
Estimation of the ability of the ADNEX model and subjective assessment to classify adnexal masses as benign or malignant when detected in patients aged 20 or under (Sensitivity, Specificity, positive predictive value, and negative predictive value) | Outcome based on histology for group 1 or follow-up for group 2 (maximum 12 months after recruitment)
  Sensitivity, Specificity, positive predictive value, and negative predictive value. Providing 95% confidence intervals and ,for ADNEX, Using several cut-offs on the risk of malignancy. Analysis will be done twice: for subgroup 1 and for subgroups 1 and 2 combined.
Estimation of the ability of the ADNEX model to predict individual risk of malignancy of adnexal masses when detected in patients aged 20 or under (Calibration) | Outcome based on histology for group 1 or follow-up for group 2 (maximum 12 months after recruitment)
  O:E ratio, and generate a flexible calibration curve. Analysis will be done twice: for subgroup 1 and for subgroups 1 and 2 combined.
Estimation of the ability of the Benign Descriptors to detect malignancies in patients aged 20 or under. | Outcome based on histology for group 1 or follow-up for group 2 (maximum 12 months after recruitment)
  Number and percentage of patients that fit any BD, only BD1, only BD2, only BD3, and only BD4 and percentage of malignancies among patients that fit any BD, only BD1, only BD2, only BD3, only BD4. We provide 95% confidence intervals for every result.
Estimation of the ability of the ADNEX model without CA125 to discriminate between benign and malignant adnexal masses when detected in patients aged 20 or under (AUC) | Outcome based on histology for group 1 or follow-up for group 2 (maximum 12 months after recruitment)
  Area under the receiver operating characteristic curve (AUC). This will be done using the estimated probability of malignancy, which equals 1 minus the estimated probability of a benign tumor. 95% confidence intervals provided. Analysis will be done twice: for subgroup 1 and for subgroups 1 and 2 combined.

SECONDARY OUTCOMES:
Occurrence of complications during follow up. | The occurrence of complications will be reported at two specific time points: at 3 months and 12 months after recruitment.
  We calculated the follow-up time from the recruitment visit until surgery, spontaneous resolution or death. If none of these events was observed, follow-up time was censored at the time of the last visit. We constructed cumulative incidence curves, considering the competing risk setting (three possible events). We report the estimated cumulative incidence of each event (with 95% confidence intervals) at 3 and 12 months of follow-up.
Examination of natural history | Initial visit, 6-8 week visit, 3-month visit, and 12-month visit.
  We will describe ultrasound characteristics (median, IQR and range for continuous variables, frequency and proportion for categorical variables) at every visit (initial visit, 6-8 week visit, 3 month visit, 12 month visit).
  This will be done overall and separately for three subgroups.
  * Patients in group 1. It does not matter whether surgery eventually took place or not.
  * Patients in group 2, and for which the mass has spontaneously resolved at the next visit (this subgroup is not applicable at the 12 month visit).
  * Patients in group 2 (this subgroup is not applicable at the 12 month visit) Exceptions: decision to operate, but it did not happen; LFU after that visit.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium